CLINICAL TRIAL: NCT06064877
Title: A Multicenter, Randomized, Double Blind, Placebo - Controlled, Phase 3 Study of Ficlatuzumab in Combination With Cetuximab in Participants With Recurrent or Metastatic (R/M) HPV -Negative Head and Neck Squamous Cell Carcinoma. (FIERCE-HN)
Brief Title: A Study of Ficlatuzumab in Combination With Cetuximab in Participants With Recurrent or Metastatic (R/M) HPV Negative Head and Neck Squamous Cell Carcinoma
Acronym: FIERCE-HN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AV-299-23-301
Record Dates: First submitted 2023-09-14; First posted 2023-10-03 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Head-and-neck Squamous-cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma
Keywords: Recurrent; Metastatic; HPV-negative; Head and Neck; Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Recurrence; Neoplasm Metastasis; Carcinoma, Squamous Cell | interventions — ficlatuzumab; Cetuximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind, Placebo-Controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Investigational Arm: ficlatuzumab plus cetuximab) (Experimental): Intravenous (IV) ficlatuzumab dose A on Day 1 (D1) and D15 of each 28-day cycle IV cetuximab on D1 and D15 of each 28-day cycle
  Interventions: Biological: Ficlatuzumab; Biological: Cetuximab
- Arm 2 (Investigational Arm: ficlatuzumab plus cetuximab) (Experimental): IV ficlatuzumab dose B on D1 and D15 of each 28-day cycle IV cetuximab on D1 and D15 of each 28-day cycle
  Interventions: Biological: Ficlatuzumab; Biological: Cetuximab
- Arm 3 (Comparator Arm: placebo plus cetuximab) (Placebo Comparator): IV placebo (saline, ficlatuzumab-matched) on D1 and D15 of each 28-day cycle IV cetuximab on D1 and D15 of each 28-day cycle
  Interventions: Biological: Cetuximab; Other: Placebo

INTERVENTIONS:
Biological: Ficlatuzumab — Ficlatuzumab (AV-299) is a humanized hepatocyte growth factor (HGF) inhibitory immunoglobulin G1 (IgG1) monoclonal antibody (mAb).
  Other Names: AV-299
  Arms: Arm 1 (Investigational Arm: ficlatuzumab plus cetuximab); Arm 2 (Investigational Arm: ficlatuzumab plus cetuximab)
Biological: Cetuximab — Cetuximab is an epidermal growth factor receptor (EGFR) antagonist.
  Other Names: Erbitux
Other: Placebo — Placebo for this study will be normal saline
  Arms: Arm 3 (Comparator Arm: placebo plus cetuximab)

SUMMARY:
The purpose of this study is to compare the efficacy and safety of ficlatuzumab plus cetuximab compared to placebo plus cetuximab in participants with recurrent/metastatic (R/M) HPV-negative Head and Neck Cancer.

The primary hypothesis is that ficlatuzumab combined with cetuximab is superior to cetuximab alone in terms of progression-free survival and/or overall survival.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled Phase 3 study is designed to compare the efficacy and safety of two dose levels of ficlatuzumab combined with cetuximab (Arm 1 or Arm 2) to a control arm of placebo plus cetuximab (Arm 3) in participants with R/M human papilloma virus (HPV)-negative HNSCC. Eligible participants must have failed prior therapy with an anti-PD-1 [programmed cell death protein 1] or PD-L1 [programmed death ligand 1] immune checkpoint inhibitor (ICI) and with platinum-based chemotherapy, administered in combination or sequentially. Failure of prior treatment may be due to progression of disease or intolerance to treatment. It is anticipated that the study will enroll approximately 410 participants across 3 arms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and ≥ 18 years of age
* Histologically and/or cytologically confirmed primary diagnosis of R/M HNSCC
* Participants with oropharyngeal cancer will be required to have proof of p16 negative status submitted on the basis of a pathology report
* At least 1 measurable lesion by contrast CT or MRI scan according to RECIST v.1.1. Such lesions must not have been previously irradiated; if the measurable lesion(s) has been irradiated, clear progression must be documented
* Participants must have failed prior therapy with an anti-PD-1/PD-L1 ICI and with platinum-based chemotherapy administered in combination or sequentially, in either the locally advanced or R/M setting. Failure of prior treatment may be due to progression of disease or intolerance to treatment
* Patient's tumor must be considered inoperable and incurable
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 with a life expectancy of at least 12 weeks
* For women of childbearing potential (WOCBP), documentation of negative serum pregnancy test within 30 days of randomization
* For WOCBP and male participants whose sexual partners are of childbearing potential, agreement to use an effective method of contraception during the study and for at least 5 months after the last dose of study treatment. Birth control methods which may be considered highly effective include methods that achieve a failure rate of less than 1% per year when used consistently and correctly.
* Ability to give written informed consent and comply with protocol requirements
* Patients with feeding tubes are eligible for the study.
* Archived tissue sample must be submitted to the Sponsor-designated laboratory within 60 days of randomization for c-Met analysis (if a tissue sample is not available, a fresh biopsy may be required prior to enrollment)

Exclusion Criteria:

* Participants who have received > 2 prior lines of anticancer therapy or prior treatment with cetuximab/alternative EGFR inhibitors for the treatment of R/M HNSCC
* History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational agent or cetuximab
* Known or suspected untreated and uncontrolled brain metastases or leptomeningeal carcinomatosis Note: Participants with locally treated brain metastases are eligible provided 2 weeks have elapsed since local therapy. Participants are allowed to continue steroid taper during the start of study treatment.
* Prior treatment with any other investigational drug or biologic agent or radiation therapy before a washout has been completed (must be completed prior to randomization):

  1. 2 weeks (14 days) or 5 half-lives, whichever is shorter, for chemotherapeutic agents, small molecules, and checkpoint inhibitors
  2. 3 weeks (21 days) or 5 half-lives, whichever is shorter, for antibody-drug conjugates
  3. 4 weeks (28 days) for cell therapies
  4. 2 weeks (14 days) for radiation therapy
* Any unresolved and significant toxicity (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] version 5.0) Grade > 2 from previous anticancer therapy (including radiation therapy), other than alopecia
* Significant cardiovascular disease, including: Cardiac failure New York Heart Association class III or IV; Myocardial infarction, severe or unstable angina within 6 months prior to randomization; History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation)
* Any other medical condition or psychiatric condition that, in the opinion of the Investigator, might interfere with the participant's involvement in the study or interfere with the interpretation of study results
* History of prior malignancy within 2 years prior to randomization (except for adequately treated non-melanoma skin cancer, carcinoma in situ of the breast or cervix, superficial bladder cancer, or early-stage prostate cancer, without evidence of recurrence; participants may or may not be on maintenance therapy)
* Participants who are positive for HBV or HCV with indication of acute or chronic hepatitis (as defined in protocol)
* Radiographic evidence (historical or at screening) of interstitial lung disease or idiopathic pulmonary fibrosis
* Female participants who are pregnant or breastfeeding

A full list of inclusion and exclusion criteria can be found in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy by overall survival of ficlatuzumab plus cetuximab vs placebo plus cetuximab in participants with recurrent/metastatic (R/M) head and neck squamous cell carcinoma (HNSCC) | From Randomization until death from any cause (Approximately 44 months)
  Overall survival (OS), defined as the time from the date of randomization to the date of death for any cause

SECONDARY OUTCOMES:
To evaluate progression-free survival (PFS) for ficlatuzumab plus cetuximab vs placebo plus cetuximab in participants with R/M HNSCC | From Randomization until disease progression or death (Approximately 44 months)
  Progression-free survival (PFS), defined as the time from randomization to the first documented progressive disease (PD) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, or death from any cause, whichever occurs first
To evaluate additional objective response rate for ficlatuzumab plus cetuximab vs placebo plus cetuximab in participants with R/M HNSCC | From Cycle 1 Day 1 until last response assessment (response assessments are every 8 weeks for the first year, every 12 weeks for years 2 and 3 and then every 6 months)
  Objective response rate (ORR), defined as the percentage of participants who have a complete response (CR) or a partial response (PR) per RECIST v1.1
To evaluate disease control rate (DCR) for ficlatuzumab plus cetuximab vs placebo plus cetuximab in participants with R/M HNSCC | From Cycle 1 Day 1 until last response assessment (response assessments are every 8 weeks for the first year, every 12 weeks for years 2 and 3 and then every 6 months)
  Disease control rate (DCR), defined for participants who have achieved a CR, PR or stable disease for at least 8 weeks per RECIST v1.1
To evaluate duration of response (DOR) for ficlatuzumab plus cetuximab vs placebo plus cetuximab in participants with R/M HNSCC | From Cycle 1 Day 1 until last response assessment (response assessments are every 8 weeks for the first year, every 12 weeks for years 2 and 3 and then every 6 months)
  Duration of response (DOR), defined as the time from first documented evidence of a confirmed CR or PR per RECIST v1.1
To compare the safety and tolerability of ficlatuzumab plus cetuximab vs placebo plus cetuximab in participants with R/M HNSCC | From Screening until 30 days after last dose
  Number of times participants experience Adverse Events (AE) or abnormal laboratory values.
To evaluate the pharmacokinetics (PK) of ficlatuzumab | From Baseline (Cycle 1 Day 1 pre-dose) until End of Treatment (Approximately 44 months)
  Serum samples will be assessed for concentrations of ficlatuzumab
To assess the immunogenicity of ficlatuzumab via antidrug antibodies (ADAs) | From Baseline (Cycle 1 Day 1 pre-dose) until End of Treatment (Approximately 44 months)
  Serum samples will be assessed for the presence of ADA to ficlatuzumab.
To assess the immunogenicity of ficlatuzumab via neutralizing antibodies (nAB) | From Baseline (Cycle 1 Day 1 pre-dose) until End of Treatment (Approximately 44 months)
  Serum samples that test positive for the presence of ADA to ficlatuzumab will be further tested for the presence of nAB.
To evaluate the quality of life (QOL) of ficlatuzumab plus cetuximab vs placebo plus cetuximab in participants with R/M HNSCC | From Baseline (Cycle 1 Day 1 pre-dose) until End of Treatment (Approximately 44 months)
  Change from baseline in overall health status and time to clinically meaningful deterioration based on scoring of standardized participant questionnaires

CONTACTS AND LOCATIONS:
Locations (110):
- United States (26):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - University of California Los Angeles, Westwood, Los Angeles, California
  - Yale School of Medicine - Smilow Cancer Hospital, New Haven, Connecticut
  - The George Washington University, Washington D.C., District of Columbia
  - AdventHealth Medical Group Oncology & Hematology at Orlando, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - MaineHealth Institute for Research, South Portland, Maine
  - University of Maryland, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Siteman Cancer Center - Washington University, St Louis, Missouri
  - Northwell Health Cancer Institute, Lake Success, New York
  - Manhattan Eye, Ear & Throat Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati - UC Health Barrett Cancer Center, Cincinnati, Ohio
  - Ohio State University, James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Oncology Consultants, Houston, Texas
  - VCU Massey Cancer Center, Richmond, Virginia
  - Medical College of Wisconsin - Froedtert Hospital Cancer Center, Milwaukee, Wisconsin
- Australia (4):
  - St George Hospital, Kogarah, New South Wales
  - St. Vincent's Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - St. John of God Murdoch Hospital, Murdoch, Western Australia
- Belgium (3):
  - CHU Liège, Liège
  - CHU Universite Catholique de Louvain, Namur
  - Vitaz-Sint-Niklaas Moerland, Sint-Niklaas
- University Hospital, Panagyurishte, Bulgaria
- Canada (5):
  - Tom Baker Cancer Centre (Alberta Health Services), Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Center - University Health Network, Toronto, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
- Czechia (5):
  - Fakultni nemocnice Brno, Brno
  - Masaryk Memorial Cancer Institute, Brno
  - Fakultni Nemocnice Olomouc, Olomouc
  - Fakultni Nemocnice Kralovske Vinohrady, Prague
  - Fakultni nemocnice Bulovka, Prague
- France (7):
  - Clinique Pasteur - Lanroze- Centre Finistérien de Radiothérapie et d'Oncologie, Brest
  - Pôle Santé Léonard de Vinci, Chambray-lès-Tours
  - Centre Léon Bérard, Lyon
  - Assistance Publique Hopitaux de Marseille (APHM)-Hôpital La Timone, Marseille
  - Institut Curie, Paris
  - Hôpital Privé des Côtes d'Armor, Plérin
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Charite-Universitaetsmedizin Berlin - Campus Virchow-Klinikum (CVK) - Medizinische Klinik mit Schwerpunkt Haematologie, Onkologie und Tumorimmunologie, Berlin
  - UNIVERSITÄTSKLINIKUM FREIBURG, Klinik für Innere Medizin I, Schwerpunkt Hämatologie, Onkologie und Stammzelltransplantation, Freiburg im Breisgau
  - Ludwig-Maximilians University, Munich
- Hungary (5):
  - Orszagos Onkologiai Intezet, Budapest
  - Petz Aladar Country Teaching Hospital, Győr
  - Josa Andras Oktatokorhaz, Nyíregyháza
  - University of Pecs - Oncology, Pécs
  - Szent Lázár Megyei Kórház, Salgótarján
- Italy (10):
  - IRCCS Istituto Scienze Neurologiche, Bologna
  - AOU Careggi, Florence
  - IRCCS Istituto Clinico Humanitas - Cancer center, Milan
  - IRCCS Ospedale San Raffaele Milano, Milan
  - Fondazione IRCCS - Istituto Nazionale Tumori - Oncologia, Milan
  - Azienda Ospedaliera Universitaria Maggiore Della Carita Novara, Novara
  - Istituto Oncologico Veneto, Padua
  - IRCCS - ICS Maugeri, Pavia
  - Universita degli Studi di Pavia - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Netherlands (2):
  - Antoni van Leeuwenhoek, Amsterdam
  - Radboud University Medical Center, Nijmegen
- Poland (2):
  - Centrum Onkologii im. prof. F. Lukaszczyka w Bydgoszczy, Bydgoszcz
  - National Research Institute of Oncology, Gliwice
- Romania (2):
  - Medisprof Cancer Center, Cluj-Napoca
  - Centrul radioterapie Amethyst Cluj-Napoca, Floreşti
- Serbia (3):
  - Institute of Oncology and Radiology of Serbia, Belgrade
  - Institute for Oncology Vojvodina, Kamenitz
  - University Clinical Center Kragujevac, Kragujevac
- South Korea (7):
  - Keimyung University Dongsan Hospital, Daegu
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Ajou University Hospital, Suwon
- Spain (12):
  - Hospital Universitario Vinalopo, Alicante
  - Institut Catala d'Oncologia - Hospital Duran i Reynals, Badalona
  - UOMI Cancer Center-Clinica Tres Torres, Barcelona
  - Institut Catala d'Oncologia (ICO) - Hospitalet, Barcelona
  - Vall d'Hebron Institut d'Oncologia (VHIO), Barcelona
  - Hospital universitario Jerez, Cadiz
  - Hospital Universitario La Paz, Madrid
  - Grupo Hospital de Madrid (HM) - Hospital Universitario Madrid Sanchinarro - Centro Integral Oncologico Clara Campal (CIOCC), Madrid
  - Hospital Universitario de Torrejón, Madrid
  - Hospital Quironsalud Malaga, Málaga
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clinico Universitario de Valencia (CHUV), Valencia
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital - Kaohsiung, Kaohsiung City
  - China Medical University Hospital (CMUH), Taichung
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan District
- United Kingdom (6):
  - NHS Grampian - Aberdeen Royal Infirmary, Aberdeen
  - The Royal Marsden NHS Foundation Trust, London
  - Sarah Cannon Research Institute, London
  - City Hospital Nottingham, Nottingham
  - The Royal Marden Hospital, Surrey, Sutton
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: No